CLINICAL TRIAL: NCT03855774
Title: Polymorphisms, Caffeine and Sleep Disorders
Acronym: SOCAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherche Biomedicale des Armees (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PDH-1-SMO-2-0509-op1; IDRCB (Other: 017-A00234-49)
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Polymorphism; Sleep Disorder; Coffee-Workers' Disease
Keywords: healthy subject; epidemiological
MeSH Terms: conditions — Sleep Wake Disorders | interventions — Polymorphism, Genetic

STUDY DESIGN:
Intervention Model Description: Epidemiological and genetic screening of a population
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Polymorphisms (Other): Classification of sleep disorders prevalence through polymorphisms
  Interventions: Genetic: Polymorphisms

INTERVENTIONS:
Genetic: Polymorphisms — Classification of sleep disorders using 22 genetic polymorphisms

SUMMARY:
Screening of a population of volunteer workers recruited on the occasion of their occupational health visit, within the Ministry of Defense and civil enterprises.

The voluntary subjects included will, after signing a consent, take a saliva sample (Kit Oragen DNA OG500) and fill out a computerized questionnaire.

A posteriori, the genotyping polymorphisms may be associated with variations in the pharmacokinetics or pharmacodynamics of caffeine will be achieved.

The primary objective is to determine whether polymorphisms (alone or in combination) of genes associated with the pharmacokinetics or pharmacodynamics of caffeine are independent risk factors for sleep disorders.

The secondary objectives are to determine the frequency of these polymorphisms and to evaluate the consequences of these associations on sleep habits (sleep time, chronotype, quality of sleep), daytime sleepiness, caffeine consumption, antecedents of accidents at work or traffic, drug consumption ...

DETAILED DESCRIPTION:
Coffee is one of the most consumed drinks in the world and its consumption has doubled in 20 years. Because of the health benefits of caffeine (present in many foods and medicines), but also adverse effects, its physiological actions deserve to be better known and its use better framed.

Indeed, caffeine is the most used psychoactive substance to prevent the deterioration of the cognitive performance of night workers and soldiers in operation. Its "strategic" use is even recommended in many armies. In its sustained-release dosage form (Caffeine 300 mg), it is the only drug, increasing alertness, authorized in the French military. Caffeine also has beneficial effects on inflammatory response, muscle activity, insulin sensitivity, cardiovascular risk, weight gain, neuroprotection, chronic pain. Usual consumption of 2 to 3 coffees a day is recommended by the American Nutrition Society.

However, coffee consumption is associated with many side effects such as anxiety, sleep disorders, increased blood pressure, cardiovascular and obstetric conditions or depression. Many authors therefore recommend limiting its use. In particular, it is considered a risk factor for sleep disorders such as insomnia.

The physiological effects and sensitivity to side effects of caffeine are characterized by very high individual variability3 related to age, sex, habitual coffee consumption, smoking, but also to genetic polymorphisms. Indeed, multiple polymorphisms are associated with changes in pharmacokinetics (see Table 1) or pharmacodynamics (efficacy, see Table 2) of caffeine. Sensitivity to caffeine is associated in particular with greater vulnerability to sleep deprivation, sleep disorders and stress.n particular, polymorphisms of the adenosine receptor (ADORA) gene, a therapeutic target for caffeine, are particularly involved in the individual variability of caffeine sensitivity, side effects and consumption habits. But many other polymorphisms of genes encoding enzymes involved in metabolism or physiological effects are also associated with the individual variability of caffeine.

On the other hand, some gene polymorphisms such as the adenosine deaminase gene (ADA) which degrades caffeine and regulates intra- and extracellular concentrations, are associated with greater vulnerability to sleep deprivation, without the effects on caffeine sensitivity are known.

Currently, it is difficult to assess the impact of these polymorphisms on the beneficial effects and / or risks associated with caffeine consumption due to their number and lifestyle, including coffee consumption. In other words, are sleep disorders favored by polymorphism and / or habitual consumption of caffeine? Are there profiles of high vulnerability to sleep deprivation and sensitivity to caffeine? Do these polymorphisms have a link with burnout, work stress, diseases?

ELIGIBILITY:
Inclusion Criteria:

* active workers

Exclusion Criteria:

* inactive subject (unemployed, student...)
* involuntary subject

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1100 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Polymorphisms and sleep disorders | 1 salivary sample (screening)
  Sleep disorders frequency by genetic polymorphism

SECONDARY OUTCOMES:
Sleep duration | 1 salivary sample (screening)
  Total sleep time (hours) in function of polymorphisms

CONTACTS AND LOCATIONS:
Locations (1):
- Fabien SAUVET, Brétigny-sur-Orge, France

IPD SHARING:
Plan to Share IPD: No